CLINICAL TRIAL: NCT00721331
Title: A Phase I, Single-Center, Randomized, Vehicle-Controlled Study to Assess the Safety and Tolerability of Topical CRx-197 Formulations in Healthy Volunteers
Brief Title: A Phase I Study to Assess the Safety and Tolerability of Topical CRx-197 Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: James Keane, Sr. Clinical Project Manager, CombinatoRx, Inc.
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CRx-197-001; EudraCT # 2008-000611-15
Record Dates: First submitted 2008-07-21; First posted 2008-07-24 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Atopic Dermatitis
Keywords: CombinatoRx; Atopic; Dermatitis; Topical; CRx-197; Normal Healthy Volunteers
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — Nortriptyline; Loratadine; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CRx-197 high dose (0.1% nortriptyline HCl + 0.3% loratadine) (Experimental)
  Interventions: Drug: nortriptyline HCl + loratadine
- CRx-197 low dose (0.1% nortriptyline HCl + 0.1% loratadine) (Experimental)
  Interventions: Drug: nortriptyline HCl + loratadine
- 0.1% nortriptyline HCl (Experimental)
  Interventions: Drug: nortriptyline HCl
- 0.1% mometasone furoate (Active Comparator)
  Interventions: Drug: mometasone furoate
- Active ingredient free vehicle cream of CRx-197 (Placebo Comparator)
  Interventions: Drug: Active ingredient free vehicle cream of CRx-197

INTERVENTIONS:
Drug: nortriptyline HCl + loratadine — Topical
  Arms: CRx-197 high dose (0.1% nortriptyline HCl + 0.3% loratadine)
Drug: nortriptyline HCl + loratadine — Topical
  Arms: CRx-197 low dose (0.1% nortriptyline HCl + 0.1% loratadine)
Drug: nortriptyline HCl — Topical
  Arms: 0.1% nortriptyline HCl
Drug: mometasone furoate — Topical
  Arms: 0.1% mometasone furoate
Drug: Active ingredient free vehicle cream of CRx-197 — Topical
  Arms: Active ingredient free vehicle cream of CRx-197

SUMMARY:
This will be a phase I, single center, randomized, vehicle-controlled, blinded study comparing two dosage strengths of CRx-197 cream, nortriptyline, an active comparator (0.1% mometasone) and placebo (the active ingredient free vehicle cream of CRx-197)in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and date the written Informed Consent prior to any study specific procedures
* Subject must be 18 to 60 years of age
* Subject must have healthy skin on which reddening can be easily recognized in the area where they will place the test fields
* Subject must be free from a condition/disease that the investigator feels interferes with the interpretation of the study results.
* Females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective medically accepted contraceptive regimen. A highly effective method of birth control is defined as those which result in a lower failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner.

Exclusion Criteria:

* Suntan, hyper- or hypo-pigmentation, or tattoos in the area where they will place the test fields
* Dark skinned persons whose skin color prevents ready assessment of skin reactions
* Cardiac disease, including recent myocardial infarction, any degree of heart block or other cardiac arrhythmias and valvular heart disease
* Mania
* Narrow angle glaucoma
* Hyperthyroidism by medical history, TSH less than LLN, or subject receiving any thyroid medication
* Severe liver disease - ALT laboratory value that exceeds 1.5x ULN
* Inflammatory dermatoses (e.g., atopic dermatoses/eczema, psoriasis)
* Any skin condition involving the test fields including but not limited to bacterial, viral, or fungal skin infections, acne, rosacea
* Active varicella, tuberculosis, syphilis or post-vaccine reactions
* Autoimmune disease (e.g., lupus erythematosis)
* Known allergic reactions or hypersensitivity to any of the components of the study treatments
* Allergy to adhesives on the patches used for occlusion in the study
* UV therapy or significant UV exposure in the four weeks before treatment application
* History of malignancy (except for treated or excised basal cell carcinoma)
* Surgery within the previous 3 months (except for minor cosmetic or dental procedures)
* History of drug or alcohol abuse (as defined by the Investigator)
* Symptoms of a clinically significant illness in the four weeks before treatment application that may influence the outcome of the study
* Positive for HIV antibody
* Systemic treatments in the four weeks prior to treatment application that may interact with any of the study drugs, such as: Glucocorticoids, MAO inhibitors, anti-depressants, anti-seizure medications, anti-psychotics and anti-histamines
* Subjects who require medications that inhibit the CYP450 2D6 pathway such as:Quinidine, Cimetidine, Type 1 anti-arrhythmic, Phenothiazines, Selective serotonin reuptake inhibitors, Reserpine, other anticholinergic drugs, and sympathomimetic drugs
* Treatment with any investigational agent within one month before treatment application for this trial
* Female subject who is pregnant , lactating, or with a positive pregnancy test
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment
* Subject is institutionalized because of legal or regulatory order

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CRx-197 as assessed by treatment emergent adverse events, physical exams, vital signs, concomitant medications/procedures and subject assessment of pruritus. | 2 months

SECONDARY OUTCOMES:
Difference in change from baseline in psoriatic infiltrate measured by ultrasound between CRx-197, nortriptyline, active comparator as well as vehicle of CRx-197 and untreated test field(s) | Days 8, 15, 22, 29 and 43
Difference in change from baseline in erythema measured by chronometry between CRx-197, nortriptyline, active comparator, vehicle of CRx-197, untreated test field(s) and normal skin | Days 8, 15, 22, 29 and 43
Modified PASI between CRx-197, nortriptyline, active comparator, vehicle of CRx-197, untreated test field(s) | Baseline, and Days 8, 15, 22, 29 and 43

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Harten, MD, Principal Investigator — Proinnovera GmbH
Locations (1):
- PROINNOVERA GmbH, Münster, Germany